CLINICAL TRIAL: NCT07075887
Title: Optic Nerve Head Evaluation Through Multimodal Blood Flow Analysis: a Prospective Observational, Multi-center Study
Acronym: FlowONH
Status: Not yet recruiting | Type: Observational
Sponsor: Barboni (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); ASST Fatebenefratelli Sacco (Other)
Responsible Party: Sponsor-Investigator, Barboni, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: FlowONH
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Neuro-Ophthalmology; Optic Neuropathies; Optic Atrophy, Hereditary, Leber; Optic Neuropathy, Anterior Ischemic; Optic Disc Drusen; Normal Tension Glaucoma (NTG)
Keywords: oct-a; ecocolordoppler; optic neuropathies
MeSH Terms: conditions — Optic Nerve Diseases; Optic Atrophy, Hereditary, Leber; Optic Neuropathy, Ischemic; Optic Disk Drusen; Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient affected by Optic Neuropathies: patients affected by acute ONH edema (NAION, papilledema, optic neuritis) patients affected by acute pseudoedema (LHON) patients affected by chronic pseudoedema (LHON, ODD) patients affected by chronic ONH neuropathies (NTG, DOA, WS) non-affected eyes in each optic neuropathy patient

SUMMARY:
OCT-A and eco-colordoppler are technologies which enable optic nerve head (ONH) blood perfusion detection. The aim of the study is to assess ONH vascular and structural components in optic neuropathies with and without ONH edema or pseudo-edema with OCT-A, and analyze ONH blood-flow with eco-colordoppler.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE The vascular component of the ONH, like that of the retina, is an essential part for the ONH homeostasis, but is considered difficult to be precisely analyzed, especially in optic nerve pathologies. Little is known about the vascular component and its role in both acute and chronic ONH diseases, particularly in conditions that cause swelling, where it is mandatory to differentiate edema from pseudo-edema.

Today, the gold standard for the vascular imaging of the retina is angiography, using either fluorescein or indocyanine green. However, conventional angiography has the disadvantage that the invasive administration of dye into the venous system is required, leading to low but potentially life-threatening side effects as allergic reactions; furthermore, data obtained are not standardizable or exploitable for a quantitative analysis. However, new technologies such as OCT-A can provide standardizable and quantifiable data on vascular structures that can be used in a statistical analysis. Additionally, eco-colordoppler ultrasound provides direct measurements of ONH blood-flow.

OBJECTIVES AND ENDPOINTS Objectives Endpoints: The aim of the study is to assess ONH vascular and structural components optic neuropathies with and without ONH edema or pseudo-edema through OCT-A (OCT-angiography) and ocular blood-flow through eco-colordoppler.

Primary Objective: to identify parameters correlated to the development and progression (prognostic biomarkers) of the diseases.

Primary Endpoint: Analysis of data collected in symptomatic and asymptomatic eyes, obtained through OCT-A in order to evaluate the relationship between functional and structural parameters in order to identify parameters correlated to the development and progression of the diseases.

Timepoint: 24 months from the enrollment.

Secondary Objectives: To assess and compare different ONH vascular components through OCT-A and eco-colordoppler in order to identify parameters correlated to the diseases.

Secondary Endpoints: To detect OCT-A parameters (vessel density, perfusion density), and eco-colordoppler parameters of central retina artery (CRA) and short posterior ciliary artery (SPCA) (systolic and diastolic flow and resistance). in order to evaluate their relationship in each optic neuropathy.

Timepoint: 24 months from the enrollment.

STUDY DESIGN OCT-A and eco-colordoppler are technologies which enable optic nerve head (ONH) blood perfusion detection. The aim of the study is to assess ONH vascular and structural components in patients affected by ONH edema or pseudo-edema with OCT-A and, in a subset of 35 patients, analyze the ONH vascular blood flow through eco-colordoppler analysis.

This is a national, prospective observational, multicentre study:

- in the cohort study (70 patients) will be included patients with chronic optic neuropathies with or without ONH pseudo-edema (NTG, ODD, DOA, WS) and contralateral eye (not affected) for each optic neuropathy and patients with acute optic neuropathies with ONH edema and pseudo-edema (NAION, LHON, papilledema, anterior neuritis). The study includes an observational period of 24 months, from baseline (date of signing of informed consent) to 24 months (4 follow-up visits 6 months apart, as in clinical practice).

Moreover, a normative database will be created in order to compare data for different ages.

Only variables obtained according to routine clinical practice, available in the hospital charts or patient's clinical records, and collected according to the study objectives can and should be documented in this study.

All patients enrolled will undergo at the same procedures reported in Figure 1, according to routine clinical practice.

In details, for every patient belonging to each disease group, a complete neuro-ophthalmologic evaluation and the data of the methodic, at baseline and in every time-point, will be collected from all the recruiting centers. Finally, the data obtained will be statistically analyzed, with the primary objective of finding a possible diagnostic and prognostic biomarker for every disease group.

The data obtained using the Orion OCT analysis Software, Voxeleron, will be analyzed by IRCCS San Raffaele.

Eco-colordoppler will be performed and analyzed at IRCCS San Raffaele, O.U. of Ophthalmology in a subset of 35 non-consecutive patients for the secondary endpoint.

Study duration Duration of enrollment: 12 months Duration of treatment: 24 months Duration of total follow-up: 24 months Duration of total study period: 36 months

STUDY POPULATION Study Participants The study will include 70 subjects, regardless of age, gender, comorbidities or drugs taken.

Inclusion Criteria

1. Participant (or parents/legal representative/tutor for minors) is willing and able to give informed consent for participation in the study;
2. patients affected by acute ONH edema (NAION, papilledema, optic neuritis);
3. patients affected by acute pseudoedema (LHON);
4. patients affected by chronic pseudoedema (LHON, ODD);
5. patients affected by chronic ONH neuropathies (NTG, DOA, WS) non-affected eyes in each optic neuropathy patient;
6. The medical product is the standard of care for the patient or the participant is taking the medicinal product according to clinical practice.

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. any other ONH disease or neurological /retinal diseases impairing the evaluation of the ONH;
2. evidence of media opacities affecting the quality of the vascular assessment;
3. patients affected Alzheimer/Parkinson disease will be considered separately.

Screening Failures Screen failures are defined as participants who consent to participate in the clinical study but do not meet the criteria for participation in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants. Minimal information includes demography, screening failure details, eligibility criteria.

No re-screening procedure is foreseen.

STUDY OBJECTIVES The aim of the study is to asses ONH vascular and structural components optic neuropathies with and without ONH edema or pseudo-edema with OCT-A and analyze the ONH vascular blood-flow with eco-colordoppler ultrasound.

The primary objective is to assess ONH vascular and structural components in optic neuropathies with and without ONH edema or pseudo-edema, through OCT-A (OCT-angiography) in order to identify parameters correlated to the diseases and obtain diagnostic and prognostic biomarkers.

The secondary objective is to evaluate ONH vascular supply using two different devices, OCT-A and eco-colordoppler, which specifically evaluate the ONH ocular and retro-ocular vessels in order to identify different disease patterns. The eco-colordoppler measurements will be collected on 35 patients enrolled only.

In accordance to the inclusion/exclusion criteria, patients to be enrolled will be those with Acute optic neuropathies with ONH edema and pseudo-edema (NAION, LHON, papilledema, anterior neuritis) and chronic optic neuropathies with or without ONH pseudo-edema (NTG, ODD, DOA, WS) and contralateral eye (not affected) for each optic neuropathy.

In the prospective observational part of the study, data will be collected from patient chart review, as is the case for clinical practice, from ICF collection up to 24 months.

For OCT-A, the following devices are allowed:

1. DRI OCT Triton, 3D Optical Coherence Tomography (Topcon Healthcare, Tokyo, Japan); OCT-A is a non-invasive imaging technique based on optical coherence tomography (OCT) developed to image and visualize vascular networks in the human retina;
2. Cirrus OCT-A (Carl Zeiss Meditech Inc., Dublin, CA, USA): OCT-A is a non-invasive imaging technique based on OCT developed to image and visualize vascular networks in the human retina;
3. Spectralis OCT (Heidelberg Engineering, Heidelberg, Germany): OCT-A is a non-invasive imaging technique based on optical coherence tomography (OCT) developed to image and visualize vascular networks in the human retina;

   The medical devices are CE marked and are used according to the indications of use of the marketing authorization released by the national Regulatory Authority (CE marking documents that the medical device complies with applicable EU legislation are required) and already used in OSR and in the other Clinical Units as part of normal clinical practice.

   Furthermore, only variables obtained according to routine clinical practice, available in the hospital charts or patient's clinical records, and collected according to the study objectives can and should be documented in this study.

   During the observational period, assessments are routinely performed in accordance with current guidelines and local standard of care. The decision of any treatment (or interruption) related to the disease under study and to concomitant diseases, is the responsibility of the treating physician and is not regulated by this protocol.

   The additional examination, eco-color doppler, in a subset of 35 patients will be performed. Eco-colordoppler is a non-invasive method developed to visualize blood flow in color and the main blood vessels. Venous blood is shown in blue, while oxygen-rich arterial blood, is displayed in red. The device used is Digital Color Doppler Ultrasound System (Sonoscape Medical Corporation), a medical device with CE mark and used according to the indications of use of the marketing authorization released by the national Regulatory Authority. The exam will be performed in every follow-up visit (6 months) at San Raffaele Hospital; the duration of the exam is about 5 minutes for each eye.

   Study object description OCT and OCT-A: structural and vascular analysis of the optic nerve head employing a coherent light to assess the morphology and vascular supply of the area (DRI OCT Triton, 3D Optical Coherence Tomography (Topcon Healthcare, Tokyo, Japan; Cirrus OCT-A (Carl Zeiss Meditech Inc., Dublin, CA, USA; Spectralis OCT (Heidelberg Engineering, Heidelberg, Germany). All the devices are equivalent in terms of results for this study. The OCT/OCT-A scans take approximately 5-10 minutes to be performed and it is not invasive.

   Ecocolordoppler: vascular assessment of the retrobulbar vessels which supply the optic nerve employing ecosonography (Digital Color Doppler Ultrasound System (Sonoscape Medical Corporation)). The exam takes 10-15 minutes and it is not invasive.

   STUDY PROCEDURES Informed Consent Informed consent is a process that is initiated prior to the individual's agreeing to participate in the study and continues throughout the individual's study participation. Consent forms will be EC-approved, and the participant will be asked to read and review the document. The investigator (according to applicable regulatory requirements) or a person designated by the investigator, and under the investigator's responsibility, will explain the research study to the participant and answer any questions that may arise. A verbal explanation will be provided in terms suited to the participant's comprehension of the purposes, procedures, and potential risks of the study and of their rights as research participants. Participants will have the opportunity to carefully review the written consent form and ask questions prior to signing. The participants should have the opportunity to discuss the study with their family or surrogates or think about it prior to agreeing to participate. The participant MUST sign the informed consent document prior to any procedures being done specifically for the study/any data is collected. Participants must be informed that participation is voluntary and that they may withdraw from the study at any time, without prejudice. A copy of the informed consent document will be given to the participants for their records. The informed consent process will be conducted and documented in the source document (including the date), and the form signed, before the participant undergoes any study-specific procedure/ any data is collected. The rights and welfare of the participants will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study.

   By providing informed consent, the patient confirms that he/she has been informed about the study and agrees to pseudonymous data collection.

   Subject Recruitment and Screening In according to inclusion/exclusion criteria will be enrolled patients (or parents/legal representative/tutor for minors) who is willing and able to give informed consent for participation in the study, affected by acute and chronic ONH neuropathies, regardless of age, gender, comorbidities or drugs taken.

   Will be included 70 patients. The enrollment will be competitive. Participants will be identified by qualified research staff, delegated for the conduction of this study. This may be done through a review of medical records, external referrals or using databases.

   The screening requirements that will be evaluated during the baseline visit are:
   * medical history/current medical history to evaluated the diagnosis in according to the inclusion criteria;
   * ophthalmological assessments (including imaging) as per routine clinical practice, to avoid the inclusion of patients with any other ONH disease or neurological /retinal that compromises ONH assessment, evidence of medial opacities that compromise the quality of vascular assessment, and/or suffering from Alzheimer's disease.

   Subject Identification Starting from the signature of the informed consent by the patient or patient's legal tutor, the subjects is considered enrolled in the clinical study.

   A subject identification code will be assigned consecutively (FLO_XXX_YYY; where FLO is the abbreviation of the Protocol Identifier, XXX is the abbreviation of the study site , YYY is the progressive subject number in increasing order starting from 001).

   A patient identification list will be kept.

   Baseline Assessments Written informed consent for participation in the study must be obtained before performing any study-related procedures (including screening evaluations). Informed Consent Forms for enrolled patients will be maintained at the study site.

   All evaluations must be completed and reviewed to confirm that patients meet all eligibility criteria before enrolment.

   The assessments will be conducted are:
   * demographics data collection;
   * data collection of medical history including clinically significant diseases, chronic and ongoing conditions surgeries, cancer history, reproductive status, and smoking history;
   * prior and concomitant medication data collection;
   * vital signs collection, as for clinical practice;
   * eco-colordoppler, (nb: performed only in OSR for 35 patients from recruiting centers)
   * ophthalmological assessments as for clinical practice: • refraction and BCVA assessed on ETDRS chart at a starting distance of 4 meters;

     • visual field test: an exam used to detect changes in peripheral vision;

     • IOP (intraocular pressure) performed prior to dilating eyes;

     • slit lamp examination;

     • dilated binocular indirect ophthalmoscopy;
     * OCT, Optical coherence tomography: is a non-invasive imaging test that use light waves to take cross-sectional pictures of your retina;
     * OCT-A, Optical coherence tomography angiography (DRI OCT Triton, 3D OCT, Topcon Healthcare, Cirrus OCT-A, Zeiss and Spectralis OCT Heidelberg): a non-invasive imaging technique based on OCT developed to image and visualize vascular networks in the human posterior pole.
   * Safety assessments: monitoring and recording adverse events, including serious adverse events and any event deemed critical to the safety of the patient.

   Visits and Follow Up The study involves 4 follow-up visits every 6 months from baseline to 24 months performed as for clinical practice.

   Ocular assessments will include the following, to be performed on both eyes at timepoints specified in the schedules of activities:

   - demographics data collection;
   * data collection of medical history including clinically significant diseases, chronic and ongoing conditions surgeries, cancer history, reproductive status, and smoking history;
   * prior and concomitant medication data collection;
   * vital signs collection, as for clinical practice;
   * eco-colordoppler, (only for the 35-patients subset);
   * ophthalmological assessments as for clinical practice:

     • refraction and BCVA assessed on ETDRS chart at a starting distance of 4 meters;

     • visual field test: an exam used to detect changes in peripheral vision;

     • IOP (intraocular pressure) performed prior to dilating eyes;

     • slit lamp examination;

     • dilated binocular indirect ophthalmoscopy;

     • OCT, optical coherence tomography: is a non-invasive imaging test that use light waves to take cross-section pictures of your retina;

     • OCT-A, optical coherence tomography angiography (DRI OCT Triton, 3D OCT, Topcon Healthcare; Cirrus OCT-A, Carl Zeiss Meditech Inc; Spectralis OCT Heidelberg Engineering): a non-invasive imaging technique based on OCT developed to image and visualize vascular networks in the human posterior pole.
   * Safety assessments: monitoring and recording adverse events, including serious adverse events and any event deemed critical to the safety of the patient.

   All assessments are captured within the specified visit window (+/-30 days).

   Definition of End of Study According to the study design, the end of the study is defined as the date on which the last patient completes the last visit (Months 24 ±30 days).

   The end of study (EoS) is defined as the date when the last patient enrolled completes their last visit (LPLV).

   Premature termination or suspension of a study This study may be temporarily suspended or prematurely terminated by the authorized Sponsor representative or the PI at any site if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to study participants, investigator, funding agency and regulatory authorities. If the study is prematurely terminated or suspended, the PI will promptly inform study participants, the EC and will provide the reason(s) for the termination or suspension. Study participants will be contacted, as applicable, and informed of changes to study visit schedule and necessary medical support.

   Circumstances that may warrant termination or suspension include, but are not limited to:

   - data that are not sufficiently complete and/or evaluable.

   In terminating the study, the Sponsor and the Principal Investigator will assure that adequate consideration is given to the protection of the subjects' interests.

   DISCONTINUATION AND WITHDRAWAL Participants are free to withdraw from participation in the study at any time upon request.

   In addition, the Investigator may discontinue or withdrawal a participant from the study for the following reason:
   * significant non-compliance with study requirements;
   * patient's decision. The reason for participant discontinuation or withdrawal from the study will be recorded on the clinical records and in Case Report Form (CRF). Subjects who sign the informed consent form and subsequently withdraw, or are withdrawn or discontinued from the study, will be replaced.

   PATIENT SAFETY All procedures in the protocol will be performed as in clinical practice; furthermore, no enrolled subjects will be exposed to an additional risk.

   The ecocolordoppler will be performed in a subset of patients (35) and its application is connected with no side effects for patients.

   STATISTICS The statistical hypotheses and the statistical methodology that will be applied to the analysis of the collected data are a fundamental component of a clinical research protocol.

   Description of Statistical Methods In the first phase, the results of the considered cohort will be analyzed from an exploratory perspective. Standard descriptive statistics, including frequencies, percentages, means, and medians, will be calculated to assess the distribution of the key study variables, previously listed in the objectives, differentiating patients based on different pathologies. Chi-square test statistics, Fisher's exact test, and Wilcoxon sum test statistics will be used as appropriate to check for differences or trends.

   The second part of the analysis will describe the results of the applied logistic models. Attention will focus on the odds ratio (OR) for the outcome of interest. The variables included in the logistic model refer to the variables detected through the tools used for perfusion pattern evaluation.

   For longitudinal analysis, mixed models will be used as they take into account correlations between repeated measures of the same individual over time.

   Sample Size Determination To obtain the study population, being in the presence of rare diseases, the sample size is based on the feasibility of recruiting individuals. However, for the statistical analysis that will be performed, it was considered that statistical tests will be significant with an alpha level of 0.05 and a beta error of 0.2.

   The total number of individuals who will be enrolled is 70 patients, of whom 15 have NAION, 15 NTG, 10 with LHON, 10 with papilledema, 5 with anterior neuropathy, 10 with ODD and 5 patients affected by DOA and WS.

   Consequently, the ONH perfusion patterns of 70 eyes will be analyzed by OCT-A and about 35 eyes by eco-colordoppler.

   Analysis Populations The analysis of data for the study will be performed when the final follow-up visit of the last patient has occurred. The data will be analyzed by IRCCS San Raffaele and, using the Orion OCT analysis Software, Voxeleron. The analysis software that will be used in support of this project is prototype software that extends Voxeleron's existing optic nerve head analysis. The existing software is both CE marked and FDA approved as licensed to and used in the Optos Monaco OCT device. This research version adds support for the devices employed in this study (Zeiss, Heidelberg, Topcon) enabling the vascular analysis for the primary objective.

   Multivariate analyses will be conducted to identify any complex relationships among multiple variables, providing a more complete understanding of the factors involved in our study. In particular, vascular components and RNFL thicknesses distributions in edema and pseudo-edema eyes will be evaluated through the Shapiro-Wilk test: if normally distributed an ANOVA with Bonferroni post-hoc test was performed for comparison; otherwise, the Kruskal-Wallis rank sum test with Dunn's post-hoc test. Lastly, a longitudinal analysis will go on to highlight changes in ONH perfusion patterns over time in the diseases under study.

ELIGIBILITY:
Inclusion Criteria:

* Participant (or parents/legal representative/tutor for minors) is willing and able to give informed consent for participation in the study
* patients affected by acute ONH edema (NAION, papilledema, optic neuritis)
* patients affected by acute pseudoedema (LHON)
* patients affected by chronic pseudoedema (LHON, ODD)
* patients affected by chronic ONH neuropathies (NTG, DOA, WS) non- affected eyes in each optic neuropathy patient

Exclusion Criteria:

* any other ONH disease or neurological /retinal disease impairing the evaluation of the ONH;
* evidence of media opacities affecting the quality of the vascular assessment;
* patients affected Alzheimer/Parkinson disease will be considered separately

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged ≥12 years affected with non-arteritic ischemic optic neuropathy (NAION, eye involved and not involved), normal tension glaucoma (NTG), Leber hereditary optic neuropathy (LHON symptomatic and asymptomatic patients [carriers]), anterior neuritis [papillitis], papilledema, optic disc drusen (ODD), dominant optic atrophy (DOA) and Wolfram Syndrome (WS)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Parameters correlated to the development and progression (prognostic biomarkers) of the diseases. | 24 months
  Analysis of data collected in symptomatic and asymptomatic eyes, obtained through OCT-A in order to evaluate the relationship between functional and structural parameters in order to identify parameters correlated to the development and progression of the diseases.

SECONDARY OUTCOMES:
To assess and compare different ONH vascular components through OCT-A and eco-colordoppler in order to identify parameters correlated to the diseases. | 24 Months
  To detect OCT-A parameters (vessel density, perfusion density), and eco-colordoppler parameters of central retina artery (CRA) and short posterior ciliary artery (SPCA) (systolic and diastolic flow and resistance). in order to evaluate their relationship in each optic neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Piero barboni, MD, Principal Investigator — IRCCS Ospedale San Raffaele

IPD SHARING:
Plan to Share IPD: No